CLINICAL TRIAL: NCT03709849
Title: Effectiveness and Safety of Bushen Culuan Decoction for Anovulatory Infertility：A Clinical Research of "Same Treatment for Different Diseases"
Brief Title: Effectiveness and Safety of Bushen Culuan Decoction for Anovulatory Infertility
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Dongzhimen Hospital, Beijing (Other); Beijing Obstetrics and Gynecology Hospital (Other); Beijing Hospital of Traditional Chinese Medicine (Other); Beijing First Hospital of integrated Chinese and Western Medicine (Other); Beijing Fengtai Hospital of Integrated Traditional and Western Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Z171100001017104
Record Dates: First submitted 2018-10-09; First posted 2018-10-17 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2018-08

CONDITIONS: Anovulatory Infertility; Abnormal Uterine Bleeding-Ovulatory Disorders; Polycystic Ovarian Syndrome; Hyperprolactinemia; Luteinized Unruptured Follicle Syndrome; Corpus Luteum Insufficiency; Ovarian Insufficiency
Keywords: Anovulatory Infertility; Bushen Culuan Decoction
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperprolactinemia | interventions — Clomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Intervention, dosage and frequency: drug: Bushen Culuan Decoction 13g tid and Clomiphene Citrate Tablets placebo 50mg qd; Dosage form: Bushen Culuan Decoction is dissolved medicine and Clomiphene Citrate Tablets placebo is tablets; Duration: the medicine will be taken from 5th day of a menstrual cycle, Bushen Culuan Decoction is taken for 14 days while Clomiphene Citrate Tablets placebo being taken for 5 days. Then patients stop taking the medicine until the 5th day of next menstrual cycle. If the patient doesn't have a regular menstrual cycle, the medicine will be taken from 5th day from vaginal bleeding caused by taking progesterone. Each treatment cycle contains 3 menstrual cycle. If the patient regains normal ovulation at the end of the first treatment cycle, she will reach the end of the whole treatment, and if not she will start the second treatment cycle. All treatment will be terminated after 2 treatment cycles.
  Interventions: Drug: experimental group: Bushen Culuan Decoction and Clomiphene Citrate Tablets placebo; Drug: control group: Clomiphene Citrate Tablets and Bushen Culuan Decoction placebo
- control group (Active Comparator): Intervention, dosage and frequency: drug: Clomiphene Citrate Tablets 50mg qd and Bushen Culuan Decoction placebo 13g tid; Dosage form: Clomiphene Citrate Tablets is tablet and Bushen Culuan Decoction placebo is dissolved medicine; Duration: the medicine will be taken from 5th day of a menstrual cycle, Clomiphene is taken for 5 days while Bushen Culuan Decoction placebo being taken for 14 days while. Then patients stop taking the medicine until the 5th day of next menstrual cycle. If the patient doesn't have a regular menstrual cycle, the medicine will be taken from 5th day from vaginal bleeding caused by taking progesterone. Each treatment cycle contains 3 menstrual cycle. If the patient regains normal ovulation at the end of the first treatment cycle, she will reach the end of the whole treatment, and if not she will start the second treatment cycle. All treatment will be terminated after 2 treatment cycles.
  Interventions: Drug: experimental group: Bushen Culuan Decoction and Clomiphene Citrate Tablets placebo; Drug: control group: Clomiphene Citrate Tablets and Bushen Culuan Decoction placebo

INTERVENTIONS:
Drug: experimental group: Bushen Culuan Decoction and Clomiphene Citrate Tablets placebo — the same as group description including dosage, frequency and duration
Drug: control group: Clomiphene Citrate Tablets and Bushen Culuan Decoction placebo — the same as group description including dosage, frequency and duration
  Other Names: brand name of Clomiphene Citrate Tablets: Fertilan

SUMMARY:
This study is to evaluate the effectiveness and safety of Bushen Culuan Decoction in the treatment of anovulatory infertility, including anovulatory abnormal uterine bleeding, polycystic ovarian syndrome, hyperprolactinemia, luteinized unruptured follicle syndrome, corpus luteum insufficiency and ovarian insufficiency, through a randomised, double-blinded, double-dummy, parallel positive controlled, adaptive multicenter clinical trial.

DETAILED DESCRIPTION:
Anovulation is one of the main causes of female infertility. Anovulatory infertility account for a proportion of 25-30% in whole female infertility.

In western medicine, hormone induced ovulation and assisted reproduction technology are two main ways to solve the problem and Clomiphene citrate is the first-line medication in ovulation induction. There are many side effects being reported in the treatment with modern medicine technique such as ovarian hyperstimulation syndrome, complication with uteroscope and puncture egg retrieval, low pregnancy rate with high ovulation rate, potential cancer occuring risk and offspring healthy risk.

Bushen Culuan Decoction is a traditional Chinese medicine recipe with 10 Chinese herbs including Tusizi, Yinyanghuo, Xianmao, Xuduan, Gouqizi, Nvzhenzi, Zelan, Shengpuhuang, Xiangfu and Chuanshanlong. Previous laboratory and exploratory clinical researches have proved Bushen Culuan Decoction had an exactly efficacy in treating anovulatory infertility safely.

In the first stage, the primary sample size In the study is 528. Half patients will receive Bushen Culuan Decoction and clomiphene citrate placebo, while the other half will receive clomiphene citrate tablets and Bushen Culuan Decoction placebo. When 1/3 of 528 patients complete the treatment, we will analysis the treatment efficacy of 6 diseases separately, and find which of them could be the target diseases of Bushen Culuan Decoction. Then we will modify the sample size depending on the result in first stage, and the research will only be processed in the target diseases being chosen. In the next stage, half patients will receive Bushen Culuan Decoction and clomiphene citrate placebo, while the other half will receive clomiphene citrate tablets and Bushen Culuan Decoction placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 21~40 years old;
2. Diagnosed with infertility;
3. Diagnosed with one of below diseases: anovulatory abnormal uterine bleeding, polycystic ovarian syndrome, hyperprolactinemia, luteinized unruptured follicle syndrome, corpus luteum insufficiency and ovarian insufficiency,
4. Diagnosed with TCM syndrome of kidney deficiency and blood stasis syndrome;
5. Patients who has normal sexual intercourse during treatment;
6. Voluntary to sign the informed consent.

Exclusion Criteria:

1. Infertility due to congenital physiological defect or malformation;
2. Infertility due to hereditary factors；
3. Infertility due to oviduct defect, immune factors, uterine fibroid, adenomyosis, endometriosis or hypoplasia of uterus；
4. Spouse has reproductive defects；
5. Severe abnormity of cardiovascular system, liver function, kidney function or hemopoietic system；
6. Allergy to experimental drugs

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 528 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Pregnancy Rate | Within 12 menstrual cycles from the first time that patient taking medicines. (Each cycle is 28 days)

SECONDARY OUTCOMES:
Ovulation Rate | At every ovulation phase (about day14 in a period cycle) within 3 or 6 menstrual cycles from the first time that patient taking medicines. (Each cycle is 28 days)
  If the patient participate 1 treatment cycle, the ovulation will be measured 3 menstrual cycles, and if the patient participate 2 treatment cycle, the ovulation will be measured 6 menstrual cycles.
Basal Body Temperature | At every morning within 3 or 6 menstrual cycles from the first time that patient taking medicines to the end of the treatment. (Each cycle is 28 days)
Endocrine Hormone | At the early follicle phase (day 3 in a period cycle) before the 1st cycle of the treatment and at the 7th cycle of the treatment. (Each cycle is 28 days)
  Including Follicle-Stimulating Hormone (FSH), Luteinizing Hormone (LH), Prolactin (PRL), Estradiol (E2), Progesterone(P), Testosterone (T).
Inhibin B | At the early follicle phase (day 3 in a period cycle) before the 1st cycle of the treatment and at the 7th cycle of the treatment. (Each cycle is 28 days)
Anti-Mullerian Hormone (AMH) | At the early follicle phase (day 3 in a period cycle) before the 1st cycle of the treatment and at the 7th cycle of the treatment. (Each cycle is 28 days)
Antral Follicle Count | At the early follicle phase (day 3 in a period cycle) before the 1st cycle of the treatment and at the 7th cycle of the treatment. (Each cycle is 28 days)
Volume of Uterus and Bilateral Ovaries at the Early Follicle Phase | At the early follicle phase (day 3 in a period cycle) before the 1st cycle of the treatment and at the 7th cycle of the treatment. (Each cycle is 28 days)
Thickness of Endometrium at the Early Follicle Phase | At the early follicle phase (day 3 in a period cycle) before the 1st cycle of the treatment and at the 7th cycle of the treatment. (Each cycle is 28 days)
Type of Endometrium at the Early Follicle Phase | At the early follicle phase (day 3 in a period cycle) before the 1st cycle of the treatment and at the 7th cycle of the treatment. (Each cycle is 28 days)
  The type of endometrium is measured by ultrasound. The type of endometrium contains type A, B, and C. Type A means the endometrium thickness is about 4-9mm, and there is a "trilaminar patterns" in the image. Type B means the endometrium thickness is about 9-12mm, the image shows moderate homogeneous echo. Type C means the endometrium thickness is about 10-14mm with a strong homogeneous echo. The type only represents different forms of endometrium, but not represents endometrium level or grade.
the Size of Dominant Follicle | At every ovulation phase (about day14 in a period cycle) within 3 or 6 menstrual cycles from the first time that patient taking medicines. (Each cycle is 28 days)
Peak-Systolic Flow Velocity of Uterus and Bilateral Ovaries | At the early follicle phase (day 3 in a period cycle) before the 1st cycle of the treatment and at the 7th cycle of the treatment. (Each cycle is 28 days)
Pulsatility Index of Uterus and Bilateral Ovaries | At the early follicle phase (day 3 in a period cycle) before the 1st cycle of the treatment and at the 7th cycle of the treatment. (Each cycle is 28 days)
  Pulsatility Index (PI) of Uterus and Bilateral Ovaries is the pulsatility index of uterine arteries and bilateral ovarial arteries. The normal range of uterine PI has no unified standard, but the smaller the index is, the better the endometrial receptivity is. Generally, when uterine PI<2, the endometrial receptivity will be good enough to get zygote implantation, and when uterine PI>3, the endometrial receptivity is too improper to get zygote implantation.
Resistant Index of Uterus and Bilateral Ovaries | At the early follicle phase (day 3 in a period cycle) before the 1st cycle of the treatment and at the 7th cycle of the treatment. (Each cycle is 28 days)
  Resistant Index (RI) of Uterus and Bilateral Ovaries is the resistant index of uterine arteries and bilateral ovarial arteries. The normal range of uterine RI has no unified standard, but the smaller the index is, the better the endometrial receptivity is.
Coagulation Indicator | At the early follicle phase (day 3 in a period cycle) before the 1st cycle of the treatment and at the 7th cycle of the treatment. (Each cycle is 28 days)
  Including prothrombin time, activated partial thromboplastin time, fibrinogen and thrombin time
Traditional Chinese Medicine Symptom Score | At the early follicle phase (day 3 in a period cycle) before the 1st cycle of the treatment and at the 7th cycle of the treatment. (Each cycle is 28 days)
  Traditional Chinese Medicine Symptom Score (point) including:
  amenorrhea (0-3); delayed menstruation (0-3); scant menstruation (0-3); weakness in lower back, waist and knees (0-3); dizziness and tinnitus (0-3); sexual apathy (0-3); fatigue (0-3); colorless transparent urination(0-3); frequent urination at night (0-3); feeling obstruction with menstruation (0-3); profuse menstruation with dark color (0-3); clot in menstruation (0-3); stabbing pain in lower abdomen area, may aggravating with sexual intercourse (0-3); dysmenorrhea (0-3) The total score will be measured by summing the subitems' score above, and the total score range is 0-42. The higher the score is, the worse the situation is.

CONTACTS AND LOCATIONS:
Overall Officials: Kun Ma, Dr., Principal Investigator — Xiyuan Hospital of China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ma K, Shi Y, He J, Teng X, Wang R, Wang G, Yu Y, Chen Y, Gong L, Yuan Y, Zhang H, Yuan B, Zhang C. The effect of Bushen Culuan Decoction on anovulatory infertile women among 6 different diseases: a study protocol for a randomized, double-blinded, positively controlled, adaptive multicenter clinical trial. Trials. 2022 Jul 8;23(1):563. doi: 10.1186/s13063-022-06289-7. PMID 35804385